CLINICAL TRIAL: NCT03989804
Title: Long-term Effects of Targeted Follow-up of New Fitness Center Members: a Blinded Randomized Controlled Trial
Brief Title: Effects of Targeted Follow-up of New Fitness Center Members
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: LR12062019
Record Dates: First submitted 2019-06-14; First posted 2019-06-18 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: New Members of Fitness Centers
Keywords: Fitness center; Physical activity; Follow-up; Members; Visits; Membership terminations; Training advisors
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Targeted follow-up (Experimental)
  Interventions: Behavioral: Targeted follow-up
- Usual practice (No Intervention): Usual practice at the fitness center is self-directed use

INTERVENTIONS:
Behavioral: Targeted follow-up — 2 phone calls and 1 e-mail delivered over 6-8 weeks after enrollment aiming to help and support members to get started using the fitness center and its services.
  Arms: Targeted follow-up

SUMMARY:
Objective: To investigate the long-term effects of targeted follow-up of new fitness center members compared to usual practice, on frequency of visits and membership terminations after four years.

Design and setting: A participant and provider blinded parallel group randomized controlled trial conducted at eight Fitness Centers in Trondheim, Central Norway.

Participants: The inclusion criteria were new members >16 years who between September 1st to 9th 2014 signed up for an ordinary contract with a minimum duration of 12 months.

Intervention: The intervention consisted of two phone calls and one e-mail delivered over 6-8 weeks after enrollment, aiming to motivate members to get started using the fitness center and its services. Usual practice at the fitness center is self-directed use.

ELIGIBILITY:
Inclusion Criteria:

* The study included new members (16 years in 2014 or older) on ordinary contracts with a minimum duration of 12 months and monthly automatic membership renewal that enrolled independent of the study at one of eight 3T-Fitness Centers in Trondheim between September 1st and September 9th, 2014.

Exclusion Criteria:

* Exclusion criteria were members with free contracts, employee contracts, cash membership, shorter membership contracts (duration <12 months) and loyalty contracts (indicates that the member is improving his old contract and is not a new member).

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Number of days with visits at the fitness center chain | 4 years
Rate of membership terminations | 4 years

SECONDARY OUTCOMES:
Number bookings to training advisors | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Siri Forsmo, PhD Prof, Study Director — Norwegian University of Science and Technology NTNU

IPD SHARING:
Plan to Share IPD: No